CLINICAL TRIAL: NCT06855160
Title: A Phase 3a, Open-Label, Randomized, Controlled Study to Evaluate the Immunogenicity and Safety of Intramuscular Administration of an Investigational Varicella Vaccine and Priorix Compared With Subcutaneous Administration of Varivax and Priorix, When Given as a First Dose to Healthy Children 12 to 15 Months of Age
Brief Title: A Study on the Immune Response and Safety of an Investigational Chickenpox Vaccine and a Marketed Measles, Mumps and Rubella Vaccine When Administered as Intramuscular Injection to Healthy Children 12 to 15 Months of Age
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 223105; 2024-518840-18-00 (Other: EU CT Number)
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Chickenpox
Keywords: Chicken pox; Candidate l varicella vaccine (VNS); Varicella; Varivax; Healthy Children
MeSH Terms: conditions — Chickenpox | interventions — Measles-Mumps-Rubella Vaccine; Hepatitis A Vaccines; Pneumococcal Vaccines

STUDY DESIGN:
Masking Description: This is an Open Label study.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- VNS+ MMR Vaccine (Experimental): Participants receive 1 dose of the candidate varicella vaccine (VNS vaccine), 1 dose of a measles, mumps, and rubella (MMR) vaccine, 1 dose of a hepatitis A virus (HAV vaccine), and 1 dose of PCV (either PCV 13 or Vaxneuvance or PCV 20) on Day 1.
  Interventions: Biological: Candidate varicella vaccine; Biological: MMR vaccine; Biological: Hepatitis A vaccine; Biological: PCV (pneumococcal conjugate vaccine) 13; Biological: PCV 20; Biological: Vaxneuvance
- VV+MMR Vaccine (Active Comparator): Participants receive 1 dose of a Marketed varicella vaccine (VV), 1 dose of a MMR vaccine, 1 dose of a HAV vaccine, and 1 dose of PCV (either PCV 13 or Vaxneuvance or PCV 20) on Day 1.
  Interventions: Biological: Marketed varicella vaccine; Biological: MMR vaccine; Biological: Hepatitis A vaccine; Biological: PCV (pneumococcal conjugate vaccine) 13; Biological: PCV 20; Biological: Vaxneuvance

INTERVENTIONS:
Biological: Candidate varicella vaccine — Investigational varicella vaccine administered intramuscularly.
  Arms: VNS+ MMR Vaccine
Biological: Marketed varicella vaccine — Marketed varicella vaccine administered subcutaneously.
  Arms: VV+MMR Vaccine
Biological: MMR vaccine — MMR vaccine administered subcutaneously or intramuscularly.
Biological: Hepatitis A vaccine — Hepatitis A vaccine co-administered intramuscularly.
Biological: PCV (pneumococcal conjugate vaccine) 13 — The 13-valent pneumococcal conjugate vaccine co-administered intramuscularly. In some countries PCV will only be administered depending on the availability, country's registration status and national recommendations for pneumococcal vaccination at the time of study conduct.
Biological: PCV 20 — The 20-valent pneumococcal conjugate vaccine co-administered intramuscularly. In some countries PCV will only be administered depending on the availability, country's registration status and national recommendations for pneumococcal vaccination at the time of study conduct.
Biological: Vaxneuvance — The Vaxneuvance (15-valent pneumococcal conjugate vaccine) co-administered intramuscularly. In some countries Vaxneuvancewill only be administered depending on the availability, country's registration status and national recommendations for pneumococcal vaccination at the time of study conduct.

SUMMARY:
This study aims to assess the immune response and safety of GSK's candidate chickenpox and marketed MMR vaccines when given to children 12 to 15 months of age via a muscle injection. It compares the GSK vaccines to Merck's chickenpox vaccine, administered just under the skin. Additionally, the study will evaluate the immune response and safety of giving the GSK vaccines along with other childhood vaccines through a muscle injection.

ELIGIBILITY:
Inclusion Criteria:

* Participant's parent(s)/ Legally acceptable representatives (LAR[s]), who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g., completion of the eDiaries, return for follow-up visits).
* Written or witnessed/thumb printed informed consent obtained from the participant's parent(s)/LAR(s) prior to performance of any study-specific procedure.
* Healthy participants as established by medical history and clinical examination before entering into the study.
* A male or female between, and including, 12 to 15 months of age (i.e., from the day of 1-year birthday until the day before 16 months of age) at the time of the administration of study interventions.
* Only for children in countries where PCV is recommended at 12 to 15 months of age as per national immunization schedule and provided as part of the study interventions:

  * Participant who previously received the primary series of PCV in the first year of life with last dose at least 60 days prior to the administration of study intervention.

Exclusion Criteria:

* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study interventions including hypersensitivity to neomycin or gelatin.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* Hypersensitivity to latex.
* Major congenital defects, as assessed by the investigator.
* Recurrent history of uncontrolled neurological disorders or seizures.
* History of measles, mumps, rubella, or varicella disease.
* Active untreated tuberculosis.
* Participants with bleeding disorders (e.g., thrombocytopenia or any coagulation disorder).
* Condition that in the judgment of the investigator would make intramuscular injection unsafe.
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study.

Prior/Concomitant therapy

* Use of any investigational or non-registered product (drug, vaccine or invasive medical device) other than the study interventions during the period beginning 30 days before the dose of study interventions administration (Day -29 to Day 1), or their planned use during the study period.
* Chronic administration of immune-modifying drugs (defined as more than 14 consecutive days in total) and/or planned use of long-acting immune modifying treatments at any time up to the end of the study.

  - Up to 90 days prior to the study intervention administration:
* For corticosteroids, this will mean prednisone equivalent >=0.5 mg/kg/day with maximum of 20 mg/day for pediatric participants. Inhaled and topical steroids are allowed.
* Administration of immunoglobulins and/or any blood products or plasma derivatives.

  - Up to 180 days prior to study interventions administration: long acting immune-modifying drugs including among others immunotherapy (e.g., tumor necrosis factor-inhibitors), monoclonal antibodies (except the ones not interfering with the immune response to the study vaccines, e.g., nirsevimab), antitumoral medication.
* Previous vaccination against measles, mumps, and rubella.
* Previous vaccination against varicella virus.
* Previous vaccination against hepatitis A virus.
* Only for children in countries where PCV is recommended at 12 to 15 months of age as per national immunization schedule and provided as part of the study interventions, participant who previously received a booster dose of any PCV.

Prior/Concurrent clinical study experience

• Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational intervention (drug/invasive medical device).

Other exclusion criteria

* Any study personnel or their immediate dependents, family, or household members.
* Child in care.
* Participants with the following high-risk individuals in their household: • Immunocompromised individuals.
* Pregnant women without documented history of varicella.
* Newborn infants of mothers without documented history of varicella.
* Newborn infants born <28 weeks of gestation

Ages: 12 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 900 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2026-09-10 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with seroresponse to Varicella Zoster Virus (VZV) anti- glycoprotein E (gE) Immunoglobulin (IgG) | At Day 43
  The seroresponse rate is defined as the percentage of participants for whom the post-vaccination Day 43 anti VZV gE IgG concentration is above the seroresponse threshold.
Geometric Mean Concentration (GMC) of anti-VZV gE IgG | At Day 43
  Concentrations of anti-VZV gE IgG are presented as GMC and expressed in milli-international units per milliliter (mIU/mL) for each group.
Percentage of participants with seroresponse to MMR antigens | At Day 43
  The seroresponse rate is defined as the percentage of participants for whom the post-vaccination Day 43 anti-measles, mumps, and rubella antibody concentrations are above the seroresponse threshold.
GMC of Anti-measles antibodies | At Day 43
GMC of Anti-mumps antibodies | At Day 43
GMC of Anti-rubella antibodies | At Day 43

SECONDARY OUTCOMES:
Percentage of participants with seroresponse to demonstrate an acceptable immune response for IM administration of MMR vaccine | At Day 43
Percentage of participants with seroresponse to MMR antigens with a reduced non-inferiority margin | At Day 43
Percentage of participants reporting each solicited administration site events post-dose of investigational VNS vaccine or VV administration | Day 1 (post-dose) to Day 4
  Solicited administration site events include injection site redness, pain, and swelling.
Percentage of participants reporting each solicited administration site events post-dose of MMR vaccine administration | Day 1 (post-dose) to Day 4
  Solicited administration site events include injection site redness, pain and swelling.
Percentage of participants reporting each solicited systemic events post-dose of study interventions administration | Day 1 (post-dose) to Day 15
  Solicited systemic events include drowsiness, loss of appetite and irritability.
Percentage of participants reporting each solicited systemic event in terms of fever post-dose of study interventions administration | Day 1 (post-dose) to Day 22
  Fever is defined as temperature greater than or equal (>=) 38.0 degrees Celsius (°C) regardless of the location of measurement (the preferred location for measuring temperature is the axilla).
Percentage of participants reporting each solicited administration site events post-dose of study interventions administration | Day 1 (post-dose) to Day 43
  Solicited administration site events include injection site varicella-like rash.
Percentage of participants reporting each solicited systemic events post-dose of study interventions administration | Day 1 (post-dose) to Day 43
  Solicited systemic events includes varicella-like rash (non-injection site), measles/rubella-like rash, and general rash (not varicella like and not measles/rubella-like).
Percentage of participants reporting unsolicited Adverse Events (AEs) post-dose of study interventions administration | Day 1 (post-dose) to Day 43
  Unsolicited AEs include any AE reported in addition to solicited events during the study, or any "solicited" symptoms with onset outside of the specified period of follow-up for solicited symptoms, are assessed for each group after the administration of all vaccines. Unsolicited AEs include nonserious and serious AEs.
Percentage of participants reporting medically attended AEs (MAAE) post-dose of study interventions administration | Day 1 (post-dose) to Day 181 (Study end)
  A MAAE is an AE for which the participant received medical attention including any symptom or illness requiring hospitalization, or an emergency room visit, or visit to/by a healthcare professional.
Percentage of participants reporting Serious AEs (SAEs) post-dose of study interventions administration | Day 1 (post-dose) to Day 181 (Study end)
  A SAE is an AE which results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or other situations that are considered serious per medical or scientific judgment.

CONTACTS AND LOCATIONS:
Locations (12):
- United States (11):
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Huntington Park, California
  - GSK Investigational Site, Sherman Oaks, California
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, Miami Lakes, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Idaho Falls, Idaho
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Lewisville, Texas
  - GSK Investigational Site, Pharr, Texas
- GSK Investigational Site, Alken, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf